CLINICAL TRIAL: NCT01366846
Title: The Persistence of Oral Tolerance Induction to Peanut and Its Immunological Basis (ITN049AD)
Brief Title: Persistence of Oral Tolerance to Peanut
Acronym: LEAP-On
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN049AD
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Results first posted 2017-01-06 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Eczema; Egg Allergy; Food Allergy; Hypersensitivity
Keywords: Peanut
MeSH Terms: conditions — Eczema; Egg Hypersensitivity; Food Hypersensitivity; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peanut avoidance after continuous peanut consumption (Experimental): These participants were the peanut consumption group of the ITN032AD (LEAP) study
  Interventions: Other: Avoidance of peanut
- Continued peanut avoidance (Experimental): These participants were the peanut avoidance group of the ITN032AD (LEAP) study
  Interventions: Other: Avoidance of peanut

INTERVENTIONS:
Other: Avoidance of peanut — All participants will be assigned to peanut avoidance as per United Kingdom (UK) public health recommendations and will avoid exposure to peanut protein during the study until the last study visit when they will receive the Oral Food Challenge.

SUMMARY:
ITN049AD (LEAP-On) Study is a continuation of the ITN032AD LEAP Study (NCT00329784).

Peanut Allergy, a recognized public health concern, is a common and potentially life-threatening food allergy for which there is no treatment. ITN032AD (LEAP) Study evaluated whether early exposure to peanut promotes tolerance and provides protection from developing peanut allergy in children who are allergic to eggs or who have severe eczema. ITN049AD (LEAP-On) Study will evaluate persistent tolerance to peanut by assessing the effect of twelve months of cessation of peanut consumption in LEAP Study participants who consumed peanut and those who avoided peanut over the previous five years.

DETAILED DESCRIPTION:
This is a two-sample comparison employing all available study participants in both arms of the LEAP (NCT00329784) study at visit 72. After obtaining informed consent, LEAP participants who are evaluable for peanut allergy at age 60 months (V60) will be enrolled into this study, the LEAP-On (NCT01366846) Study. All LEAP-On participants will avoid peanut for an additional 12 months regardless of their previous allocation to the LEAP Study consumption arm (Group A) or the LEAP Study avoidance arm (Group B).

At V72, after 12 months of this new intervention, all participants will have skin prick testing (SPT), specific IgE and a repeat oral challenge to peanut to determine the frequency of peanut allergy in both groups. The LEAP Study decision table will be used to determine the presence of peanut allergy. Briefly, peanut allergy will be based on the presence of a positive oral peanut challenge with objective signs of allergy. Tolerance will be established on the basis of a negative oral peanut challenge (tolerating 5 g of peanut protein in the absence of symptoms). For participants who do not have an oral challenge or an oral challenge at V72 with a determinate outcome, the following criteria will be used to determine their outcome at V72:

* If the participant is tolerant and has an IgE > 0.1 and/or SPT > 0 mm at V60, the participant will be considered non-evaluable and will not be included in the analysis.
* For all other participants, the V60 outcome will be applied to the V72 outcome (last observation carried forward).

Predictive values of peanut-specific IgE and/or SPT will not be used in the LEAP-On study because participants in the peanut consumption arm in the LEAP study are tolerating peanuts despite having high IgE and/or SPT.

ELIGIBILITY:
Inclusion Criteria:

* All LEAP Study participants who are evaluable for peanut allergy at year 5 by LEAP (ClinicalTrials.gov ID NCT00329784) Study criteria.
* Parent or guardian willing to provide informed consent.

Exclusion Criteria:

* Unable or unwilling to comply with study intervention and procedures.
* Participation in other food allergy intervention trials.

Ages: 5 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 556 (Actual)
Dates: Start 2011-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gideon Lack, MD, Study Chair — Evelina Children's Hospital
Locations (1):
- Evelina Children's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
ITN049AD (LEAP-On) is a continuation of the ITN032AD LEAP Study. The plan is to share data in: 1.) ImmPort, a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts; and 2.)TrialShare, a clinical trials research portal developed by the Immune Tolerance Network.

REFERENCES:
- [Background] Du Toit G, Roberts G, Sayre PH, Bahnson HT, Radulovic S, Santos AF, Brough HA, Phippard D, Basting M, Feeney M, Turcanu V, Sever ML, Gomez Lorenzo M, Plaut M, Lack G; LEAP Study Team. Randomized trial of peanut consumption in infants at risk for peanut allergy. N Engl J Med. 2015 Feb 26;372(9):803-13. doi: 10.1056/NEJMoa1414850. Epub 2015 Feb 23. PMID 25705822
- [Background] Santos AF, Du Toit G, Lack G. Is the use of epinephrine a good marker of severity of allergic reactions during oral food challenges? J Allergy Clin Immunol Pract. 2015 May-Jun;3(3):429-30. doi: 10.1016/j.jaip.2014.12.009. No abstract available. PMID 25956314
- [Background] Gruchalla RS, Sampson HA. Preventing peanut allergy through early consumption--ready for prime time? N Engl J Med. 2015 Feb 26;372(9):875-7. doi: 10.1056/NEJMe1500186. Epub 2015 Feb 23. No abstract available. PMID 25705823
- [Result] Du Toit G, Sayre PH, Roberts G, Sever ML, Lawson K, Bahnson HT, Brough HA, Santos AF, Harris KM, Radulovic S, Basting M, Turcanu V, Plaut M, Lack G; Immune Tolerance Network LEAP-On Study Team. Effect of Avoidance on Peanut Allergy after Early Peanut Consumption. N Engl J Med. 2016 Apr 14;374(15):1435-43. doi: 10.1056/NEJMoa1514209. Epub 2016 Mar 4. PMID 26942922
- See also: LEAP Study informational website — http://www.leapstudy.co.uk/
- See also: Immune Tolerance Network website — http://www.immunetolerance.org/
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- Available data/document: Individual Participant Data Set: LEAP-On (ITN049AD) — https://www.itntrialshare.org/
- Available data/document: Study protocol synopsis; datasets and figures from published NEJM 2016 article: LEAP-On (ITN049AD) — https://www.itntrialshare.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From among those who completed the LEAP study (protocol ID ITN032AD, ClinicalTrials.gov ID NCT00329784), 556 subjects were recruited between 26 May 2011 and 6 June 2014 at Evelina Children's Hospital in London, UK.
Pre-assignment Details: In the LEAP trial, participants were stratified into strata based on a peanut allergen skin prick test (SPT). Participants were either SPT negative (0mm wheal) or SPT positive (1-4 mm wheal). Participants were then randomized into treatment groups within each stratum. This configuration was preserved in LEAP-On (this trial)
Groups:
- Negative Stratum - Continued Peanut Avoidance Group: Participants who had a negative response to a peanut allergen skin prick test (no measurable wheal) and were then randomized into the peanut avoidance group for the duration of LEAP (protocol ID ITN032AD, ClinicalTrials.gov ID NCT00329784). As with participants of all treatment groups, these participants avoided peanut protein during the following LEAP-On study (this trial)
- Negative Stratum - Peanut Avoidance After Consumption Group: Participants who had a negative response to a peanut allergen skin prick test (no measurable wheal) and were then randomized into the peanut consumption group for the duration of LEAP (protocol ID ITN032AD, ClinicalTrials.gov ID NCT00329784). As with participants of all treatment groups, these participants avoided peanut protein during the following LEAP-On study (this trial).
- Positive Stratum - Continued Peanut Avoidance Group: Participants who had a positive response to a peanut allergen skin prick test (a wheal measuring between 1 and 4 mm) and were then randomized into the peanut avoidance group for the duration of LEAP (protocol ID ITN032AD, ClinicalTrials.gov ID NCT00329784). As with participants of all treatment groups, these participants avoided peanut protein during the following LEAP-On study (this trial).
- Positive Stratum - Peanut Avoidance After Peanut Consumption G: Participants who had a positive response to a peanut allergen skin prick test (a wheal measuring between 1 and 4 mm) and were then randomized into the peanut consumption group for the duration of LEAP (protocol ID ITN032AD, ClinicalTrials.gov ID NCT00329784). As with participants of all treatment groups, these participants avoided peanut protein during the following LEAP-On study (this trial).
Period: Overall Study
Arm/Group | Negative Stratum - Continued Peanut Avoidance Group | Negative Stratum - Peanut Avoidance After Consumption Group | Positive Stratum - Continued Peanut Avoidance Group | Positive Stratum - Peanut Avoidance After Peanut Consumption G
Started | 235 | 228 | 47 | 46
Completed | 232 | 224 | 46 | 45
Not Completed | 3 | 4 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Communication Difficulties | 1 | 4 | 0 | 1
Not completed — Scheduling Conflicts | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat
Groups:
- Negative Stratum - Peanut Avoidance Group: Participants who had a negative response to a skin prick test for peanut allergen (no measurable wheal) and were then randomized to the peanut avoidance group. Participants were instructed to avoid exposure to peanut protein during study participation.
- Negative Stratum - Peanut Consumption Group: Participants who had a negative response to a skin prick test for peanut allergen (no measurable wheal) and were then randomized to the peanut consumption group. Participants were fed at least 2 g of peanut protein 3 times per week (a total of 6g). The preferred peanut source was Bamba (a peanut snack), although peanut butter was an acceptable substitute. After age 3, participants were allowed to eat whole peanuts.
- Positive Stratum - Peanut Avoidance Group: Participants who had a positive response to a skin prick test for peanut allergen (a wheal measuring between 1 and 4 mm) and were then randomized to the peanut avoidance group. Participants were instructed to avoid exposure to peanut protein during study participation.
- Positive Stratum - Peanut Consumption Group: Participants who had a positive response to a skin prick test for peanut allergen (a wheal measuring between 1 and 4 mm) and were then randomized to the peanut consumption group. Participants were fed at least 2 g of peanut protein 3 times per week (a total of 6g). The preferred peanut source was Bamba (a peanut snack), although peanut butter was an acceptable substitute. After age 3, participants were allowed to eat whole peanuts.
- Total: Total of all reporting groups
Arm/Group | Negative Stratum - Peanut Avoidance Group | Negative Stratum - Peanut Consumption Group | Positive Stratum - Peanut Avoidance Group | Positive Stratum - Peanut Consumption Group | Total
Number analyzed (Participants) | 235 | 228 | 47 | 46 | 556
Age, Customized [Mean (Standard Deviation); unit: Months]
  Age in Months | 61.0 (3.44) | 61.7 (4.19) | 60.6 (3.76) | 61.4 (4.98) | 61.3 (3.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 102 | 14 | 18 | 219
  Male | 150 | 126 | 33 | 28 | 337
Region of Enrollment [Number; unit: participants]
  United Kingdom | 235 | 228 | 47 | 46 | 556

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Peanut Allergy (PA) at 72 Months of Age - by Skin Prick Test Stratum
Description: At 72 months of age, eligible participants were given an oral food challenge (oral intake of 5g of peanut protein in a single dose). Participants were considered to not have peanut allergy (PA) if they experienced no reaction following the food challenge. Those who did react were offered a double-blind, placebo-controlled food challenge with a total of 13.7g of peanut protein administered in increments. These participants were considered to have PA if they experienced a reaction at any point during the dose escalation. For participants for whom data from the oral food challenge were either inconclusive or not available, a diagnostic algorithm based on the results of a SPT and the values for peanut-specific IgE were used to determine whether or not a participant should be considered to have PA.
Time Frame: 72 months
Population: Intent-to-treat with available data at 72 months
Measure: Count of Participants; unit: Participants
Arm/Group | Negative Stratum - Peanut Avoidance Group | Negative Stratum - Peanut Consumption Group | Positive Stratum - Peanut Avoidance Group | Positive Stratum - Peanut Consumption Group
Number analyzed (Participants) | 234 | 224 | 46 | 46
Participants | 34 | 7 | 18 | 6
Statistical Analysis 1: Comparison: Negative Stratum - Peanut Avoidance Group vs Negative Stratum - Peanut Consumption Group; Comparison of the percentage of subjects with peanut allergy in the Continued Peanut Avoidance Group to that of the Peanut Avoidance After Peanut Consumption Group within the SPT-negative stratum; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Positive Stratum - Peanut Avoidance Group vs Positive Stratum - Peanut Consumption Group; Comparison of the percentage of subjects with peanut allergy in the Continued Peanut Avoidance Group to that of the Peanut Avoidance After Peanut Consumption Group within the SPT-positive stratum; Test type: Superiority or Other; p = 0.004, Chi-squared

2. Primary Outcome: Number of Participants With Peanut Allergy (PA) at 72 Months of Age - by Treatment Group
Description: At 72 months of age, eligible participants were given an oral food challenge (oral intake of 5g of peanut protein in a single dose). Participants were considered to have no peanut allergy (PA) if they experienced no reaction following the food challenge. Those who did react were offered a double-blind, placebo-controlled food challenge with a total of 13.7g of peanut protein administered in increments. These participants were considered to have PA if they experienced a reaction at any point during the dose escalation. For participants for whom data from the oral food challenge were either inconclusive or not available, a diagnostic algorithm based on the results of a SPT and the values for peanut-specific IgE were used to determine whether or not a participant should be considered to have PA.
Time Frame: 72 months
Population: Intent-to-treat with available data at 72 Months
Measure: Count of Participants; unit: Participants
Groups:
- Continued Peanut Avoidance Group: In the LEAP trial (protocol ID ITN032AD, ClinicalTrials.gov ID NCT00329784), participants assigned to the peanut avoidance group were instructed to avoid exposure to peanut protein during study participation. This group continued to avoid peanut protein throughout LEAP-On (this trial).
- Peanut Avoidance After Peanut Consumption Group: In the LEAP trial (protocol ID ITN032AD, ClinicalTrials.gov ID NCT00329784), participants assigned to the peanut consumption group were asked to consume at least 2 g of peanut protein 3 times per week (a total of 6g). The preferred peanut source was Bamba (a peanut snack), although peanut butter was an acceptable substitute. After age 3, participants were allowed to eat whole peanuts. Upon transitioning from LEAP (protocol ID ITN032AD, ClinicalTrials.gov ID NCT00329784) to LEAP-On (this trial), participants were instructed to avoid peanut protein during study participation.
Arm/Group | Continued Peanut Avoidance Group | Peanut Avoidance After Peanut Consumption Group
Number analyzed (Participants) | 280 | 270
Participants | 52 | 13
Statistical Analysis 1: Comparison: Continued Peanut Avoidance Group vs Peanut Avoidance After Peanut Consumption Group; Comparison of the percentage of participants with peanut allergy in the Continued Peanut Avoidance Group to that of the Peanut Consumption Group across both the SPT-negative and SPT-positive strata; Test type: Superiority or Other; p < 0.001, Chi-squared

3. Primary Outcome: Number of Participants With Peanut Allergy (PA) at 72 Months of Age - by Skin Prick Test Stratum in the Per Protocol Population
Description: At 72 months of age, eligible participants were given an oral food challenge (oral intake of 5g of peanut protein in a single dose Participants were considered to have no peanut allergy (PA) if they experienced no reaction following the food challenge. Those who did react were offered a double-blind, placebo-controlled food challenge with a total of 13.7g of peanut protein administered in increments. These participants were considered to have PA if they experienced a reaction at any point during the dose escalation. For participants for whom data from the oral food challenge were either inconclusive or not available, a diagnostic algorithm based on the results of a SPT and the values for peanut-specific IgE were used to determine whether or not a participant should be considered to have peanut allergy.
Time Frame: 72 months
Population: Per Protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Negative Stratum - Peanut Avoidance Group | Negative Stratum - Peanut Consumption Group | Positive Stratum - Peanut Avoidance Group | Positive Stratum - Peanut Consumption Group
Number analyzed (Participants) | 226 | 171 | 46 | 36
Participants | 34 | 7 | 18 | 6
Statistical Analysis 1: Comparison: Negative Stratum - Peanut Avoidance Group vs Negative Stratum - Peanut Consumption Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Positive Stratum - Peanut Avoidance Group vs Positive Stratum - Peanut Consumption Group; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.027, Chi-squared

4. Primary Outcome: Number of Participants With Peanut Allergy (PA) at 72 Months of Age - by Treatment Group in the Per Protocol Population
Description: At 72 months of age, eligible participants were given an oral food challenge (oral intake of 5g of peanut protein in a single dose Participants were considered to have no peanut allergy (PA) if they experienced no reaction following the food challenge. Those who did react were offered a double-blind, placebo-controlled food challenge with a total of 13.7g of peanut protein administered in increments. These participants were to have PA if they experienced a reaction at any point during the dose escalation. For participants for whom data from the oral food challenge were either inconclusive or not available, a diagnostic algorithm based on the results of a SPT and the values for peanut-specific IgE were used to determine whether or not a participant should be considered to have PA.
Time Frame: 72 months
Population: Per Protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Continued Peanut Avoidance Group | Peanut Avoidance After Peanut Consumption Group
Number analyzed (Participants) | 272 | 207
Participants | 52 | 13
Statistical Analysis 1: Comparison: Continued Peanut Avoidance Group vs Peanut Avoidance After Peanut Consumption Group; Comparison of the percentage of subjects with peanut allergy in the Continued Peanut Avoidance Group to that of the Peanut Avoidance After Peanut Consumption Group across both the SPT-negative and SPT-positive strata; Test type: Superiority or Other; p < 0.001, Chi-squared

5. Secondary Outcome: Number of Participants With Peanut Allergy (PA) at 60- and 72-month Visits Within the Peanut Avoidance After Peanut Consumption Group
Description: At 60 and 72 months of age, eligible participants were given an oral food challenge (intake of 5g of peanut protein in a single dose). Participants were considered to have no peanut allergy (PA) if they experienced no reaction following the food challenge. Those who did react were offered a double-blind, placebo-controlled food challenge with a total of 9.4g/13.7g (month 60/month 72) of peanut protein administered in increments. These participants were considered to have PA if they experienced a reaction at any point during the dose escalation. For participants for whom data from the oral food challenge were either inconclusive or not available, a diagnostic algorithm based on the results of a SPT and the values for peanut-specific IgE were used to determine whether or not a participant should be considered to have PA.
Time Frame: 60 months and 72 months
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Peanut Avoidance After Peanut Consumption Group
Number analyzed (Participants) | 270
Participants
  Month 60 | 10
  Month 72 | 13
Statistical Analysis 1: Comparison: Peanut Avoidance After Peanut Consumption Group; Comparison of the percentage of subjects with peanut allergy in the Peanut Avoidance After Peanut Consumption Group at month 60 to that of the Peanut Avoidance After Peanut Consumption Group at month 72 across both the SPT-negative and SPT-positive strata; Test type: Superiority or Other; p = 0.250, Exact McNemar

6. Secondary Outcome: Number of Peanut Avoidance After Peanut Consumption Group Participants With Peanut Allergy (PA) at 60- and 72-month Visits Within in the Per Protocol Population
Description: as for outcome 5
Time Frame: 60 months and 72 months
Population: Per Protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Peanut Avoidance After Peanut Consumption Group
Number analyzed (Participants) | 207
Participants
  Month 60 | 10
  Month 72 | 13
Statistical Analysis 1: Comparison: Peanut Avoidance After Peanut Consumption Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.250, Exact McNemar

ADVERSE EVENTS:
Time Frame: 4 years, 3 months
Description: During active follow-up study ITN049AD
Arm/Group | Negative Stratum - Peanut Avoidance Group | Negative Stratum - Peanut Consumption Group | Positive Stratum - Peanut Avoidance Group | Positive Stratum - Peanut Consumption Group
Serious Adverse Events (participants affected / at risk) | 12/235 | 7/228 | 3/47 | 2/46
Other Adverse Events (participants affected / at risk) | 206/235 | 182/228 | 45/47 | 38/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Negative Stratum - Peanut Avoidance Group (N=235) | Negative Stratum - Peanut Consumption Group (N=228) | Positive Stratum - Peanut Avoidance Group (N=47) | Positive Stratum - Peanut Consumption Group (N=46)
Anaphylactic reaction (Immune system disorders) | 2 (3) | 1 (1) | 2 (2) | 2 (2)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema infected (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Negative Stratum - Peanut Avoidance Group (N=235) | Negative Stratum - Peanut Consumption Group (N=228) | Positive Stratum - Peanut Avoidance Group (N=47) | Positive Stratum - Peanut Consumption Group (N=46)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 5 (5) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 12 (13) | 15 (18) | 4 (5) | 4 (4)
Pyrexia (General disorders) | 13 (14) | 12 (12) | 3 (3) | 3 (3)
Food allergy (Immune system disorders) | 42 (57) | 26 (42) | 16 (20) | 13 (19)
Seasonal allergy (Immune system disorders) | 12 (13) | 5 (6) | 2 (2) | 2 (2)
Ear infection (Infections and infestations) | 8 (9) | 9 (12) | 4 (4) | 2 (2)
Gastroenteritis (Infections and infestations) | 23 (26) | 12 (12) | 4 (4) | 4 (4)
Lower respiratory tract infection (Infections and infestations) | 20 (22) | 7 (8) | 2 (4) | 5 (5)
Respiratory tract infection (Infections and infestations) | 40 (54) | 39 (47) | 11 (13) | 9 (11)
Rhinitis (Infections and infestations) | 46 (52) | 41 (44) | 9 (12) | 8 (10)
Varicella (Infections and infestations) | 11 (11) | 16 (16) | 0 (0) | 4 (4)
Viral infection (Infections and infestations) | 13 (15) | 11 (11) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 3 (4) | 3 (3) | 3 (4) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 32 (41) | 20 (34) | 4 (5) | 7 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 14 (21) | 3 (4) | 5 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 18 (21) | 19 (21) | 8 (13) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 61 (79) | 42 (56) | 14 (15) | 9 (9)
Rash (Skin and subcutaneous tissue disorders) | 10 (10) | 10 (10) | 2 (2) | 3 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (5) | 13 (15) | 5 (5) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No